CLINICAL TRIAL: NCT04691856
Title: Efficacy of Intravenous Paracetamol and Ibuprofen on Postoperative Pain and Morphine Consumption in Hysterectomy: Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Efficacy of Intravenous Paracetamol and Ibuprofen on Postoperative Pain and Morphine Consumption in Hysterectomy
Acronym: ibupro-hyst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sedat Akbas, Assoc Prof, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sedatakbas7
Record Dates: First submitted 2020-12-24; First posted 2020-12-31 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain Management
Keywords: Postoperative pain; Intravenous paracetamol; Intravenous ibuprofen; Hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Analgesia, Patient-Controlled; Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Placebo-Controlled Clinical Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): 250 ml saline will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received Morphine Sulfate with intravenous patient controlled analgesia (IV PCA) pump during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml/h, lockout period: 7 min.
  Interventions: Drug: Morphine Sulfate; Drug: Morphine
- Intravenous paracetamol (Active Comparator): 1 g paracetamol will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received Morphine Sulfate with intravenous patient controlled analgesia (IV PCA) pump during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml/h, lockout period: 7 min.
  Interventions: Drug: Morphine Sulfate; Drug: Intravenous paracetamol; Drug: Morphine
- Intravenous ibuprofen (Active Comparator): 800 mg ibuprofen (diluted with 250 ml saline) will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received Morphine Sulfate with intravenous patient controlled analgesia (IV PCA) pump during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml/h, lockout period: 7 min.
  Interventions: Drug: Morphine Sulfate; Drug: Intravenous ibuprofen; Drug: Morphine

INTERVENTIONS:
Drug: Morphine Sulfate — Patients will be received morphine with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.
  Other Names: Intravenous patient-controlled analgesia
Drug: Intravenous paracetamol — 1 g paracetamol will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received morphine with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.
  Other Names: paracetamol
  Arms: Intravenous paracetamol
Drug: Intravenous ibuprofen — 800 mg ibuprofen (diluted with 250 ml saline) will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received morphine with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.
  Other Names: ibuprofen
  Arms: Intravenous ibuprofen
Drug: Morphine — All patients were instructed to use intravenous patient-controlled analgesia (IV PCA). All administrations will be applied through IV infusion over 30 minutes. Patients will be received morphine with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml, lockout period: 7 min.

SUMMARY:
To compare the effects of intravenous paracetamol and ibuprofen on postoperative pain and morphine consumption in patients undergoing hysterectomy surgery and the side effects associated with opioids.

DETAILED DESCRIPTION:
All surgical procedures are associated with acute pain and inflammation, varying degrees of severity for the patients, causing significant stres and discomfort. Effective postoperative pain management in hysterectomy can reduce complications and improve postoperative care. In postoperative pain, multimodal analgesic techniques are used to provide synergistic effects through different nociceptive mechanisms.

Hysterectomy is the second most common gynecological surgery performed after cesarean section. It is known that effective postoperative analgesia management decreases complications and increases patients' comfort.

Various analgesics are used for pain. Opioids, frequently used for postoperative pain, are the most frequently used drug group. The combination of opioids with adjuvant agents may reduce the opioid consumption used systemically. Side effects such as sedation, respiratory depression, nausea, vomiting, rash and urinary retention that develop secondary to opioids may also be reduced by the combination of supplemental analgesics.

Adjuvant agents, including nonsteroidal antiinflammatory drugs (NSAID), may be used in combination with opioids. NSAIDs do not only reduce pain, but also control the underlying inflammatory process. In addition, combining NSAIDs and opioids can help reduce the side effects by reducing administration of total opioid consumption.

Intravenous ibuprofen is the first and only intravenous NSAID approved in the United States for both pain and fever control in adults. It has been reported in multicenter, randomized, double-blind, placebo-controlled studies that IV ibuprofen is safe and effective in postoperative pain management for abdominal hysterectomy and orthopedic surgeries.

Intravenous paracetamol is an analgesic and antipyretic agent used as a first step drug for pain and fever control in adults and children. It has been clearly shown that IV paracetamol, with analgesic efficacy and safety profile, reduces analgesic requirements for pain management. It has also been shown that it provides better analgesic efficacy and reduces the opioid consumption when used in combination with opioids.

The investigators aimed to compare the effects of intravenous paracetamol and ibuprofen on postoperative pain and morphine consumption in patients undergoing hysterectomy surgery and the side effects associated with opioids.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists scores 1-3
* 18-65 years

Exclusion Criteria:

* American Society of Anesthesiologists scores IV,
* Under the age of 18,
* Over the age of 65,
* Peptic ulcer disease,
* Hepatic and renal dysfunction,
* Severe cardiovascular and pulmonary disease,
* Allergic history to propofol, fentanyl, rocuronium, paracetamol, ibuprofen and morphine,
* Emergency surgery,
* Refused informed consent form

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Hysterectomy
Enrollment: 66 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | From end of anesthesia (15 minutes after awakening of anesthesia) to postoperative 24-hour period
  Visual Analog Scale (VAS, 0-10)

SECONDARY OUTCOMES:
Sedation score | From end of anesthesia (15 minutes after awakening of anesthesia) to postoperative 24-hour period
  Ramsey sedation score (1-6)
Cumulative morphine consumption (mg) | From end of anesthesia (15 minutes after awakening of anesthesia) to postoperative 24-hour period
  All patients will be received morphine with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 100 mg morphine in 200 mL of saline (0.5 mg/ml). The PCA device was adjusted as infusion: 0 ml/h, bolus: 1 ml/h, lockout period: 7 min. Then cumulative morphine consumption will be recorded as milligram (mg).

CONTACTS AND LOCATIONS:
Overall Officials: Sedat MD AKBAS, Study Director — Inonu University Medical Faculty
Locations (1):
- Sedat Akbas, Malatya, Türkiye-Türkçe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tunali Y, Akcil EF, Dilmen OK, Tutuncu AC, Koksal GM, Akbas S, Vehid H, Yentur E. Efficacy of intravenous paracetamol and dexketoprofen on postoperative pain and morphine consumption after a lumbar disk surgery. J Neurosurg Anesthesiol. 2013 Apr;25(2):143-7. doi: 10.1097/ANA.0b013e31827464af. PMID 23360885

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT04691856/Prot_SAP_000.pdf